CLINICAL TRIAL: NCT04634448
Title: The Prevalence of Appendiceal Tumours in Patients Presenting With a Periappendicular Abscess - A Nationwide Prospective Cohort Study
Brief Title: The Prevalence of Appendiceal Tumours in Periappendicular Abscess
Acronym: PeriAPPAC-T
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Oulu University Hospital (Other); Tampere University Hospital (Other); Kuopio University Hospital (Other); Jyväskylä Central Hospital (Other); Mikkeli Central Hospital (Other); Lapland Central Hospital (Unknown); Vaasa Central Hospital, Vaasa, Finland (Other); Seinajoki Central Hospital (Other); North Karelia Central Hospital (Other); South Carelia Central Hospital (Other); Päijänne Tavastia Central Hospital (Other); Satakunta Central Hospital (Other)
Responsible Party: Principal Investigator, Paulina Salminen, Professor of Surgery, Turku University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PeriAPPAC-T
Record Dates: First submitted 2020-11-09; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Appendix Abscess; Appendicitis; Appendix Mass; Appendix Cancer; Appendix Nec; Appendix Tumor; Appendix Diseases
MeSH Terms: conditions — Appendicitis; Appendiceal Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective clinical cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interval appendectomy (Other): For all patients presenting with a periappendicular abscess, an interval appendectomy is planned at 2 to 3 months after initial conservative treatment, which is considered mandatory for all patients over 35 years of age. If a patient is under 35 and asymptomatic and does not want to undergo surgery, a follow-up MRI at 1 year will be performed.
  Interventions: Procedure: Interval appendectomy
- Follow-up MRI (Other): For all patients presenting with a periappendicular abscess, an interval appendectomy is planned at 2 to 3 months after initial conservative treatment, which is considered mandatory for all patients over 35 years of age. If a patient is under 35 and asymptomatic and does not want to undergo surgery, a follow-up MRI at 1 year will be performed.
  Interventions: Diagnostic Test: Follow-up MRI at 1 year

INTERVENTIONS:
Procedure: Interval appendectomy — interval appendectomy at 2 to 3 months after the initial non-operative treatment
  Arms: Interval appendectomy
Diagnostic Test: Follow-up MRI at 1 year — follow-up MRI at 1 year for asymptomatic patients under 35 years of age not wanting to undergo surgery
  Arms: Follow-up MRI

SUMMARY:
Complicated and uncomplicated appendicitis follow different epidemiological trends also suggesting different pathophysiology behind these two different forms of appendicitis. In 3-10% of patients complicated acute appendicitis is enclosed by formation of a circumscribed periappendicular abscess. The clinically established practice of antibiotic therapy and drainage, if necessary, has been shown safe and effective, allowing the acute inflammatory process to subside in more than 90% of cases without surgery. The need of subsequent interval appendectomy has been questioned with appendicitis recurrence risk varying between 5-26%.

During trial enrollment in our randomized Peri-APPAC trial based on the interim analysis results with 17% appendiceal tumor rate in the study population, the trial was prematurely terminated based on ethical concerns. All the follow-up group patients were re-evaluated and surgery was offered and recommended to all follow-up group patients. After this assessment and additional appendectomies, two more tumors were diagnosed resulting in neoplasm rate of 20% in the whole study group all diagnosed in patients over 40 years and the neoplasm rate in patients over 40 years was 29%.

Based on high appendiceal tumor rate in patients over 40 years, the appendiceal neoplasm rate needs to be further evaluated in prospective patient cohorts undergoing interval appendectomy as interval appendectomy is generally well tolerated and obliterates the risk of missing a possible tumor. In a recent systematic review of retrospective cohort studies with 13.244 acute appendicitis patients the overall appendiceal tumor rate was 1% after appendectomy, but in patients presenting with appendiceal inflammatory mass the neoplasm rate varied from 10% to 29%.

This nationwide prospective multicenter cohort study is designed to assess the prevalence of appendiceal tumors associated with a periappendicular abscess. All consecutive patients presenting with a periappendicular abscess are recommended to undergo interval appendectomy after initial conservative treatment with antibiotic therapy and drainage, if necessary. All patients older than 35 years will undergo laparoscopic interval appendectomy at 2 to 3 months and this is also recommended for the patients between 18 and 35 years of age. Asymptomatic patients under 35 years not willing to undergo interval appendectomy, will undergo a follow-up MRI at 1 year after the initial non-operative treatment.

DETAILED DESCRIPTION:
Complicated and uncomplicated appendicitis follow different epidemiological trends also suggesting different pathophysiology behind these two different forms of appendicitis. In 3-10% of patients complicated acute appendicitis is enclosed by formation of a circumscribed periappendicular abscess. The clinically established practice of antibiotic therapy and drainage, if necessary, has been shown safe and effective, allowing the acute inflammatory process to subside in more than 90% of cases without surgery. The need of subsequent interval appendectomy has been questioned with appendicitis recurrence risk varying between 5-26%.

During trial enrollment in our randomized Peri-APPAC trial, the high incidence of appendiceal tumors in the study population alarmed the researchers. Based on the interim analysis results with 17% appendiceal tumor rate in the study population, the trial was prematurely terminated based on ethical concerns. All the follow-up group patients were re-evaluated and surgery was offered and recommended to all follow-up group patients. After this assessment and additional appendectomies, two more tumors were diagnosed resulting in neoplasm rate of 20% in the whole study group all diagnosed in patients over 40 years and the neoplasm rate in patients over 40 years was 29%.

Based on high appendiceal tumor rate in patients over 40 years, the appendiceal neoplasm rate needs to be further evaluated in prospective patient cohorts undergoing interval appendectomy as interval appendectomy is generally well tolerated and obliterates the risk of missing a possible tumor. In a recent systematic review of retrospective cohort studies with 13.244 acute appendicitis patients the overall appendiceal tumor rate was 1% after appendectomy, but in patients presenting with appendiceal inflammatory mass the neoplasm rate varied from 10% to 29%.

This nationwide prospective multicenter cohort study is designed to assess the prevalence of appendiceal tumors associated with a periappendicular abscess. All of the study hospitals will have a common clinical protocol of recommending interval appendectomy to all patients presenting with a periappendicular abscess after initial conservative treatment with antibiotic therapy and drainage, if necessary. Considering the high rate of appendiceal neoplasms, all patients older than 35 years will undergo laparoscopic interval appendectomy at 2 to 3 months after the successful initial non-operative treatment and this is also recommended for the patients between 18 and 35 years of age. Asymptomatic patients under 35 years not willing to undergo interval appendectomy, will undergo a follow-up MRI at 1 year after the initial non-operative treatment.

ELIGIBILITY:
Inclusion Criteria:

* periappendiceal abscess proven by CT, Mri or US

Exclusion Criteria:

* patient declines to participate, complicated appendicitis without periappendiceal abscess

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
The Prevalence of Appendiceal Tumours in Periappendicular Abscess | 2-3 months (interval appendectomy)
  The Prevalence of Appendiceal Tumours in Patients Presenting With a Periappendicular Abscess - A Nationwide Prospective Cohort Study

SECONDARY OUTCOMES:
Tympanic temperature | Day 0 (on primary admission)
  All patients
Imaging (primary diagnosis) finding | Day 0 (on primary admission)
  All patients
Duration of symptoms on admission | Day 0 (on primary admission)
  All patients
Laboratory value: CRP | Day 0 (on primary admission) up to 3-5 days (discharge from the hospital)
  CRP
Laboratory value: leuckocytes | Day 0 (on primary admission) up to 3-5 days (discharge from the hospital)
  leuk
Laboratory value: neutrophils | Day 0 (on primary admission) up to 3-5 days (discharge from the hospital)
  neutr
Laboratory value: hemoglobin | Day 0 (on primary admission) up to 3-5 days (discharge from the hospital)
  Hb
Laboratory value: kreatinine | Day 0 (on primary admission) up to 3-5 days (discharge from the hospital)
  Krea
Laboratory value: CEA | Day 0 (on primary admission) up to 3-5 days (discharge from the hospital) and up to 1 year, if no interval appendectomy
  CEA
Laboratory value. Cg-A | Day 0 (on primary admission) up to 3-5 days (discharge from the hospital)and up to 1 year, if no interval appendectomy
  Cg-A
Primary nonoperative treatment | Day 0 and up to one week
  All patients, treatment details
Colonoscopy: endoscopic findings and histology | 2 weeks to 2 months prior to planned interval appendectomy
  In both intervention groups
Interval appendectomy specimen histology | At 3 months
  Interval appendectomy patients
Complications after interval appendectomy | at the time of surgery
  Clavien-Dindo classification, interval appendectomy group
Duration of hospital stay | up to 2 years
  All patients both at primary treatment, interval appendectomy and follow-up
Follow-up MRI findings | at 1 year
  In case the patient does not under interval appendectomy
follow-up CEA | at 1 year
  Follow-up MRI patients
follow-up CgA | at 1 year
  Follow-up MRI patients
Surgery after follow-up MRI | up to 10 years
  Follow-up with MRI patients

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Salminen, prof, MD, Principal Investigator — Turku University Hospital

IPD SHARING:
Plan to Share IPD: Yes
IPD is available from the PI upon request, if needed.
Supporting Information: Study Protocol, SAP
Time Frame: At study completion
Access Criteria: Please see above.

REFERENCES:
- [Derived] Salminen R, Alajaaski J, Rautio T, Hurme S, Nordstrom P, Makarainen E, Lietzen E, Pinta T, Gronroos-Korhonen M, Rantanen T, Andersen J, Mattila A, Kossi J, Riikola A, Paajanen H, Matikainen M, Pokela V, Salminen P. Appendiceal Tumor Prevalence in Patients With Periappendicular Abscess. JAMA Surg. 2025 May 1;160(5):526-534. doi: 10.1001/jamasurg.2025.0312. PMID 40172884